CLINICAL TRIAL: NCT06648343
Title: Effect of Cognitive and Physical Function Training in the Elderly
Brief Title: Intensive Home-based Complex Training in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Collaborators: Ministry of Science and ICT, Republic of Korea (Other Government); The Korea Health Technology R&D Project through the Korea Health Industry Development Institute (Unknown)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Prof, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-09-005
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Elderly
Keywords: cognitive training; physical exercise; older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Intensive cognitive and physical training
  Interventions: Other: Intensive cognitive and physical training

INTERVENTIONS:
Other: Intensive cognitive and physical training — The cognitive and physical training program consists of 25-35 minutes of cognitive training (memory, attention, visuospatial orientation) and 10-15 minutes of physical training (stretching, strength training, coordination, and aerobic exercise). Additionally, participants will be instructed to perform 30-40 minutes of aerobic exercise 3-4 times per week

SUMMARY:
This is a single-arm intervention study aimed at investigating whether a 4-week program of daily cognitive and physical activities, lasting 2-3 hours per day, produces significant changes in functional levels in healthy adults aged 65 and older.

DETAILED DESCRIPTION:
Purpose of the Clinical Study The aim of this clinical study is to evaluate the effects of cognitive and physical function training in elderly individuals (including those with subjective cognitive decline) to aid in the development of preventive and therapeutic methods for dementia.

Study Participants -Number of Participants and Basis This is a pilot study, and no formal sample size calculation was performed. The study will include 30 participants.

Clinical Study Procedure and Assessment Visit 1 (Screening) During the screening visit, the researcher will select participants based on the inclusion/exclusion criteria. All study-related assessments will take place after obtaining consent. However, if any assessments were performed within 7 days of the screening visit, those results may be used instead. The following activities will be conducted:

Visit 2 (Baseline Assessment) Baseline assessments will be conducted, and Visit 1 and Visit 2 can be performed on the same day. The following activities will be conducted:

After the baseline assessment, participants will receive self-training materials for a 4-week program, jointly developed by EBS (Korea Educational Broadcasting System) and Bundang CHA Hospital. The cognitive and physical function training program will be conducted five times a week for 40 minutes per session. The effectiveness will be evaluated through baseline assessments, and post-training assessments will be conducted after 4 weeks to analyze the results.

The cognitive and physical training program consists of 25-35 minutes of cognitive training (memory, attention, visuospatial orientation) and 10-15 minutes of physical training (stretching, strength training, coordination, and aerobic exercise). Additionally, participants will be instructed to perform 30-40 minutes of aerobic exercise 3-4 times per week.

Participants will be provided with a self-training log to record whether they performed the exercise and to check adherence.

Visit 3 (Post-training Assessment) After completing the 4-week cognitive and physical training program, post-training assessments will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older.
* Individuals capable of independent daily living (including mobility).
* Individuals who fully understand the study and voluntarily agree to participate, providing written consent.

Exclusion Criteria:

* MMSE score less than 20 (19 or below will be excluded).
* Individuals with neurological conditions such as stroke, brain tumor, cerebral palsy, dementia, or Parkinson's disease.
* Individuals with serious medical conditions (cardiovascular, gastrointestinal, respiratory, endocrine, etc.) that compromise their general health.
* Participants currently involved in other clinical studies or who participated in another clinical trial within the past 30 days.
* Any other conditions deemed inappropriate for study participation by the researcher.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
K-MMSE (Korean Mini-Mental Status Examination) | 4 weeks
  The Mini-Mental State Examination (MMSE) is a widely used screening tool for assessing cognitive function. It is designed to evaluate different cognitive abilities, including memory, attention, language, orientation, and visuospatial skills. The MMSE consists of a series of questions and tasks, with a maximum score of 30 points.

SECONDARY OUTCOMES:
RBANS (Repeatable Battery for the Assessment of Neuropsychological Status) | 4 weeks
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) is a neuropsychological test battery used to evaluate cognitive functioning across multiple domains. It is often employed to assess cognitive decline, dementia, and other conditions that affect memory and cognition. RBANS is designed to be both comprehensive and time-efficient, typically taking around 20-30 minutes to administer.
K-MBI (Korean Version of the Modified Barthel Index) | 4 weeks
  The Modified Barthel Index (MBI) is a widely used tool to measure a person's ability to perform activities of daily living (ADL) independently. It assesses functional mobility and self-care tasks, which are essential for independent living. The MBI is an adaptation of the original Barthel Index and is commonly used in rehabilitation settings to evaluate the progress of patients recovering from conditions such as stroke, brain injuries, or other impairments that affect physical function.
BBS (Berg Balance Scale) | 4 weeks
  The Berg Balance Scale (BBS) is a clinical test used to measure balance and assess the risk of falling in individuals, particularly older adults or those with neurological conditions. The test consists of 14 tasks that evaluate both static and dynamic balance, such as standing, sitting, and moving between positions. Each task is scored on a scale from 0 to 4, with a maximum total score of 56. Higher scores indicate better balance and lower fall risk.

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided